CLINICAL TRIAL: NCT02603614
Title: A Randomized, Double Blind, Placebo-Controlled, Dose Escalating, Cross Over Designed Study to Assess the Safety and Tolerability, Pharmacokinetics, and Pharmacodynamics of Open-Label, Continuous Subcutaneous Infusion of Cenderitide Via the Insulet Drug Delivery System in Chronic Stable Heart Failure Subjects With Moderate Renal Impairment
Brief Title: Safety Study of Cenderitide in Chronic Stable Heart Failure With Moderate Renal Impairment
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Capricor Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDNP-578-02
Record Dates: First submitted 2015-11-05; First posted 2015-11-13 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2018-10

CONDITIONS: Heart Failure; Renal Insufficiency
Keywords: Chronic Heart Failure; Renal Insufficiency; Natriuretic Peptides; Cenderitide
MeSH Terms: conditions — Heart Failure; Renal Insufficiency | interventions — cenderitide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cenderitide-Placebo (Experimental): Infusion Period A: Cenderitide Infusion Period B: Placebo
  This is a randomized, double-blind, placebo-controlled, cross-over trial. The sequence was either cenderitide crossed over to placebo or placebo crossed over to cenderitide, with the sequence divided into two 7-day infusion periods (Infusion Period A and Infusion Period B).
  Interventions: Drug: Cenderitide; Drug: Placebo
- Placebo-Cenderitide (Experimental): Infusion Period A: Placebo Infusion Period B: Cenderitide
  This is a randomized, double-blind, placebo-controlled, cross-over trial. The sequence was either cenderitide crossed over to placebo or placebo crossed over to cenderitide, with the sequence divided into two 7-day infusion periods (Infusion Period A and Infusion Period B).
  Interventions: Drug: Cenderitide; Drug: Placebo

INTERVENTIONS:
Drug: Cenderitide — Cenderitide is a dual receptor natriuretic peptide.
Drug: Placebo — Placebo control

SUMMARY:
CNDP-578-02 is a randomized, double-blind, placebo-controlled, dose-escalation, crossover design trial. Eight evaluable subjects (n=8) with chronic stable heart failure and moderate renal impairment will be randomized (1:1) to receive cenderitide or placebo. Enrolled subjects will begin with Infusion Period A where they will receive up to 7 days of continuous, subcutaneous, dose-escalating infusions of cenderitide or placebo via the Insulet Drug Delivery System. Enrolled subjects will then cross over into Infusion Period B where they will receive up to 7 days of continuous, subcutaneous, dose-escalating infusions of cenderitide or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent after reviewing the design and risks of the study and prior to completing any study-related procedure
* Willing and able to understand and comply with all study procedures and requirements, including in-patient stay
* Current or historical New York Heart Association (NYHA) functional class ≥ II
* Glomerular Filtration Rate (GFR) ≥ 30 and ≤ 60 mL/min at the time of screening
* Systolic blood pressure 120-160 mmHg at the time of screening
* Stable and compliant treatment with oral medications for at least 4 weeks prior to screening
* Body Mass Index (BMI) ≥18 and ≤45 kg/m2 at the time of screening
* Women of child bearing potential (WOCBP) and males must agree to use at least two forms of contraception, of which one includes a barrier method (male condom) by the male partner, during study participation and continued for at least 90 days after the conclusion of the final infusion rate. In addition, sperm donations by male subjects are not permitted during the subject's participation in the research study and for at least 90 days after the conclusion of the final infusion rate. This criterion may be waived for male subjects who have undergone a vasectomy at least 6 months prior to screening
* Willing and able to abstain from drugs, alcohol, and tobacco during study participation

Exclusion Criteria:

* Hypersensitivity or allergy to natriuretic peptides
* Acute decompensated heart failure (ADHF) within 30 days prior to randomization
* Clinical diagnosis of acute coronary syndrome (ACS) within 30 days prior to randomization
* Symptomatic postural hypotension
* Concomitant medication of an aldosterone blocker (e.g., eplerenone or spironolactone) within 30 days prior to randomization
* Potassium of ≥ 5.0 mmol/L
* Evidence of uncorrected volume or sodium ≤ 130 mmol/L within 24 hours prior to randomization
* Clinically significant aortic or mitral valve stenosis
* Acute myocarditis or hypertrophic obstructive, restrictive, or constrictive cardiomyopathy (not including restrictive mitral filling patterns)
* Significant pulmonary disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-12; Primary Completion 2016-03-31 (Actual); Study Completion 2016-03-31 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as evaluated by incidence and severity of treatment-emergent adverse events, concomitant medications, and changes from baseline in lab assessments, vital signs, physical exams, and ECGs per subject and for the study as a whole. | Evaluated throughout the duration of a subject's participation in the study until 7 days post completion of the final study infusion of cenderitide or placebo.
Pharmacokinetics of cenderitide by assessing Cmax | Pre-dose baseline, 24, 48, 72, 96, 120, 144, 168 hours after the start of the infusion period, and 4 and 24 hours post conclusion of the infusion period.
Pharmacokinetics of cenderitide by assessing tmax | Pre-dose baseline, 24, 48, 72, 96, 120, 144, 168 hours after the start of the infusion period, and 4 and 24 hours post conclusion of the infusion period.
Pharmacokinetics of cenderitide by assessing AUC(0-discharge) | Pre-dose baseline, 24, 48, 72, 96, 120, 144, 168 hours after the start of the infusion period, and 4 and 24 hours post conclusion of the infusion period.
Pharmacodynamics as assessed by observed vital signs and changes from baseline. | Evaluated throughout the duration of a subject's participation in the study until 7 days post completion of the final study infusion of cenderitide or placebo.
Pharmacodynamics as assessed by observed weight and changes from baseline. | Evaluated daily during each infusion period (Days -1 - 9)
Pharmacodynamics as assessed by daily volume difference between liquid intake and urine output (i.e., daily fluid balance) and changes from baseline. | Evaluated daily during each infusion period (Days -1 - 9)
Pharmacodynamics as assessed by observed plasma cystatin C and changes from baseline. | Pre-dose baseline, 24, 48, 72, 96, 120, 144, 168 hours after the start of the infusion period, and 4 and 24 hours post conclusion of the infusion period.
Pharmacodynamics as assessed by observed plasma cGMP and changes from baseline. | Pre-dose baseline, 24, 48, 72, 96, 120, 144, 168 hours after the start of the infusion period, and 4 and 24 hours post conclusion of the infusion period.
Pharmacodynamics as assessed by observed urinary cGMP and changes from baseline. | Evaluated daily during each infusion period (Days -1 - 9)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Ascheim, MD, Study Director — Capricor Therapeutics, Inc.
Locations (1):
- Orange County Research Center, Tustin, California, United States

IPD SHARING:
Plan to Share IPD: No